CLINICAL TRIAL: NCT03512314
Title: Open-label Extension Study with Tadekinig Alfa (r-hIL-18BP) to Monitor Safety and Tolerability in Patients with IL-18 Driven Monogenic Autoinflammatory Conditions: NLRC4 Mutation and XIAP Deficiency
Brief Title: Therapeutic Use of Tadekinig Alfa in NLRC4 Mutation and XIAP Deficiency As Open Label Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB2 Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLE-NLRC4/XIAP.2016.001
Record Dates: First submitted 2018-04-09; First posted 2018-04-30 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: XIAP Deficiency; NLRC4-MAS
MeSH Terms: conditions — Lymphoproliferative Syndrome, X-Linked, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tadekinig alfa (Experimental): Active drug treatment during 26 weeks
  Interventions: Drug: Tadekinig alfa

INTERVENTIONS:
Drug: Tadekinig alfa — Open label, 26 weeks on Tadekinig alfa treatment.
  Other Names: r-hIL-18BP

SUMMARY:
This is an open-label extension study for patients previously enrolled in the AB2 Bio Ltd. ongoing Phase III clinical trial NLRC4/XIAP.2016.001 (IND N° 127953). This OLE study will evaluate the long-term safety and tolerability of Tadekinig alfa in patients suffering from pediatric monogenic autoinflammatory diseases harboring deleterious mutations of NLRC4 and XIAP.

DETAILED DESCRIPTION:
Pediatric auto-inflammatory conditions related to spontaneous activating mutations of the NLRC4 and with recurrent MAS-like flares with constitutive IL-18 hypersecretion, may require long-term blockade of the IL-18 pathway.

Patients with X-linked inhibitor of apoptosis (XIAP) deficiency and suffering from Hemophagocytic-Lymphohistiocytosis (HLH), a MAS-like syndrome, also show high levels of serum IL-18 and may benefit from IL-18 blockade treatment until a curative hematopoietic stem cell transplantation can be performed The safety of IL-18 blockade during long-term periods is of major interest for the treatment of these patients

ELIGIBILITY:
Inclusion Criteria: (both criteria must be met)

1. Patients have participated in AB2 Bio ltd. Phase III clinical trial NLRC4/XIAP.2016.001 (IND N° 127953) by one of the following mechanisms : a) Patients that have completed the first 18-week RCT phase of the preceding clinical trial but were not eligible for the RW phase due to flare symptoms. Or b) Patients that completed the first 18-week RCT phase and completed the RW phase of the preceding clinical trial. Or c) Patients who have exited either the RCT or RW phase of the preceding clinical trial due to treatment failure requiring rescue immunosuppression. Such patients must wait a minimum of 4 weeks after treatment discontinuation from the preceding clinical trial before enrolling in this OLE. If patients do not consent to enroll in the OLE after their early termination in the main study, they will be asked to continue with the planned visits of the main study
2. Women of childbearing potential with negative urine pregnancy test (UPT) at all visits

Exclusion Criteria:

1. Patients may not enter the OLE if they voluntarily withdrew from RCT or RW study or if the time period between participation exceeds 3 months
2. Evidence or history of malignancy
3. Evidence of invasive or life-threatening infection
4. History of tuberculosis
5. Life-threatening bleeding within 2 weeks of screening
6. Vaccination with a live vaccine within the previous 3 months
7. Evidence of severe organ compromise including but not limited to: (see details in the protocol)
8. Pregnant or breastfeeding females
9. Inability to follow highly effective birth control recommendations during the study and until 1 month after the end of the treatment.
10. Inability to provide informed consent, and also assent if applicable
11. Life expectancy less than 4 weeks
12. Concomitant use of other immunosuppression except NSAIDs, glucocorticoids, cyclosporine, tacrolimus, IL-1 inhibitors (Anakinra, Canakinumab, or Rilonacept)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Reports of adverse events | 26 weeks
  The incidence, nature and severity of AEs will be reported
Reports of abnormal physical examination | 26 weeks
  Measurements will be done using the modified Auto-inflammatory Disease Activity Index (mAIDAI) including multiple measurements aggregated as 1 / 0.
Reports of abnormal laboratory results | 26 weeks
  Report of clinically significant abnormal laboratory results (i.eSerum CRP (ug/mL), Serum Ferritin (ng/mL). and any other abnormal lab results
Immunogenicity evaluation | 26 weeks
  Generation of anti-recombinant human Interleukin-18 Binding Protein (anti-rhIL-18BP) antibodies
Evaluation of the local tolerability at the injection site | 26 weeks
  Evaluation will be done based on the Local Tolerability Index where the patients will be asked to assess the degree of pain, redness, swelling, bruising, tenderness and itching, they are experiencing from each injection.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Behrens, MD, Principal Investigator — Children Hospital of Philadelphia
Locations (11):
- United States (8):
  - UCSD _ Department of Pediatrics / Rady Children's Hospital, La Jolla, California
  - Shands Children's Hospital, Gainsville, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital _ Baylor College of Medicine, Houston, Texas
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal
- Universitätsklinikum Freiburg, Centrum für Chronische Immundefizienz (CCI) - Paediatric Unit, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
This information will be provided soon